CLINICAL TRIAL: NCT05596500
Title: Influence of Vitero Supplementation (Rice-Pea-Blueberry Sport Gel Formulation) on Exercise-Induced Oxinflammation
Brief Title: Blueberry-protein Supplementation and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: SinnovaTek (Unknown); North Carolina State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 22-0013
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Response
Keywords: blueberries; exercise; inflammation
MeSH Terms: conditions — Motor Activity; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized treatment, double blinded procedures, crossover
Who Masked: Participant, Investigator
Masking Description: Investigators and study participants will be blind to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blueberry-protein gel (Experimental): Blueberry polyphenols (1 cup fresh blueberries equivalent) from extract with 20 grams rice-pea protein in a gel.
  Interventions: Dietary Supplement: Blueberry-protein gel
- Blueberry gel (Active Comparator): Blueberry polyphenols (1 cup fresh blueberries equivalent) from extract in a gel.
  Interventions: Dietary Supplement: Blueberry gel
- Placebo (Placebo Comparator): All proximate matched ingredients except for the blueberry polyphenols and plant protein.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Blueberry-protein gel — Sport gel with blueberry extract and plant protein.
  Arms: Blueberry-protein gel
Dietary Supplement: Blueberry gel — Sport gel with blueberry extract only.
  Arms: Blueberry gel
Dietary Supplement: Placebo — Sport gel without the blueberry extract polyphenols and without protein.
  Arms: Placebo

SUMMARY:
This study is the human clinical trial component of an SBIR grant with Sinnovatek (funded). Cyclists (n=20) will consume a blueberry-protein, blueberry, or placebo supplement for 2 weeks prior to cycling for 2.5 h at high intensity. Washout periods (2 weeks) will separate the 3 trials, and the cyclists will crossover (randomized) to one of the two others supplements for 2 weeks, and then engage in additional 2.5 h cycling bouts. Blood and urine samples will be collected pre- and post-supplementation for each of the 3 trials. Blood samples will also be collected immediately after and 1.5h- and 24h-post-exercise. Blood samples will be analyzed for inflammation and oxidative stress outcomes. Urine samples will be analyzed for blueberry gut-derived phenolics.

DETAILED DESCRIPTION:
PURPOSE: To investigate the influence of 2-weeks blueberry, blueberry-protein, versus placebo gel supplementation (randomized, crossover) on oxinflammation markers and blueberry gut-derived phenolics after 2.5 h intensive cycling exercise in 20 subjects.

HYPOTHESIS: We hypothesize that 2-weeks blueberry or blueberry-protein polyphenol (500 mg/day) versus placebo gel supplementation will attenuate post-exercise increases in inflammation and oxidative stress biomarkers.

RESEARCH PROCEDURES The research procedures will be conducted at the Human Performance Laboratory (Room 1201, Plants for Human Health Institute Building, 600 Laureate Way), operated by Appalachian State University at the North Carolina Research Campus (NCRC) in Kannapolis, NC. Subjects will come to the lab for orientation/baseline testing with pre-supplementation blood sample collections, three 2.5 h cycling sessions, and additional lab visits to provide 1-day 7:00 am recovery blood samples) (thus 9 total lab visits). The total amount of time subjects will be asked to volunteer for this study is about 20 hours at the Human Performance Laboratory (over a 10-week period).

Orientation/Baseline Testing (Lab Visit #1) Two weeks prior to the 2.5 h cycling session, subjects will report to the Human Performance Laboratory at approximately 7:00-8:00 am. A blood sample will be collected in an overnight fasted state to coincide with the same time of the day for the post-supplementation blood draw. Study participants will be tested for maximal aerobic capacity (VO2max) during a graded, cycle ergometer test with the Cosmed CPET metabolic device (Cosmed, Rome, Italy). Body composition will be measured with the seca BIA and Bod Pod body composition analyzer (Life Measurement, Concord, CA). Demographic and training histories will be acquired with questionnaires. Gel blueberry, blueberry protein, or placebo supplements will be supplied. 3-day food records will be supplied with thorough instructions. Participants will be given two 24-h urine collection kits with thorough written and oral instruction on collection procedures. The first 24-h urine collection bottle will be collected during the 24-h period immediately after lab visit #1 and turned in the next morning. Supplementation will start right after the urine is turned in. The second 24-h urine collection bottle will be collected during the 24-h period immediately prior to lab visit #2. Subjects will collect every drop of urine in the collection bottle for 24 hours.

2-Week Supplementation Periods Study participants will be randomized to Vitero (rice-pea-blueberry) gel, blueberry gel, and placebo gel trials, with supplements ingested daily for 2-weeks prior to participation in the first 2.5 h cycling session. After a 2-week washout period, participants will repeat all procedures two more times using the counterbalanced supplements.

Vitero (500 mg total blueberry polyphenols per day) or placebo (containing all proximate matched ingredients except for the phytoactive polyphenolics) gels will be consumed with breakfast and lunch. The gels will look identical. The placebo has been formulated in house (NCSU at the Plants for Human Health Institute).

2.5 h Cycling Session (Lab Visit #2) During the 3-day period prior to each of three the 2.5 h cycling sessions, subjects will taper exercise training and ingest a moderate-carbohydrate diet using a food list restricting high fat foods, visible fats, and polyphenols. Subjects will record all food and beverage intake during the 3-day period, with macro- and micro-nutrient intake assessed using the Food Processor dietary analysis software system (ESHA Research, Salem, OR).

Study participants will report to the Human Performance Lab in an overnight fasted state and provide a blood sample, ingest the rice-pea-blueberry, blueberry, or placebo gel with water, and then cycle 2.5h at high intensity (60% watts max) while ingesting water alone (3 ml/kg every 15 minutes). Blood samples will be collected at 0 h, 1.5 h, and 21 h post-exercise.

Testing protocol during the lab sessions with the 2.5 h cycling session:

1. 7:00 am: Provide blood sample and delayed onset of muscle soreness (DOMS) rating.
2. 7:10 am: Ingest supplements with water.
3. 7:30 am: Start 2.5 h cycling session. Subjects are to complete the 2.5 h session at an average of 60% watts max. Subjects will use their own bicycles on Saris trainers with Zwift software. A course with moderate difficulty will be utilized using the Zwift software. Heart rate and rating of perceived exertion (RPE) will be recorded every 30 minutes, and workload (watts) continuously monitored using the Zwift software system. Oxygen consumption, carbon dioxide production, respiratory exchange ratio, and ventilation will be measured using the Cosmed Quark CPET metabolic cart every 30 minutes. The total distance cycled in 2.5 h will be recorded. Subjects will consume 3 ml/kg water every 15 min. No other beverage or food containing energy or nutrients will be allowed during the cycling time sessions.
4. ~10:00 am to 11:30 am: Immediate-post-exercise, and 1.5-h recovery blood samples. Blood samples will be taken via venipuncture immediately after completing the cycling session, and then 1.5-h post-exercise. Subjects will be allowed to shower and change clothes. DOMS questionnaire will be administered immediately post-exercise and 1.5-h post-exercise. Subjects will ingest no food or beverage other than water (7 ml/kg during the 1.5 h post-exercise period). Subjects will ingest the supplement gels, and then be allowed to leave the lab. Subjects will be instructed to adhere to the food list requirements, and to keep exercise training intensity moderate.
5. 7:00 am, next morning: 21-h blood sample and DOMS rating (Lab visit #3).

Washout/Crossover/Repeat Subjects will engage in a 2-week washout period without supplements, crossover, and then repeat all procedures (Lab visits #4,5,6, and then #7,8,9).

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Ages 18-65 years.
* Non-smoker.
* Regularly compete in road races (category 1 to 5) and/or are capable of cycling 2.5 h in a laboratory setting (using their own bicycles on Saris training systems).
* Agree to train normally, maintain weight, and avoid the regular use of large-dose vitamin and mineral supplements, herbs, and medications that influence inflammation and immune function (especially Advil, Motrin, aspirin, and similar anti-inflammatory drugs) for the duration of the 6-week study. (Review supplement and medication use with the Research Manager during orientation).
* Categorized as "low risk" using the American College of Sports Medicine screening questionnaire.
* Generally healthy and without chronic disease including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 and 2 diabetes, rheumatoid arthritis.

Exclusion Criteria:

* Inability to comply with study requirements.
* Body weight below 100 pounds.
* Pregnant or breastfeeding.
* Any other concurrent condition which, in the opinion of the primary investigator (PI), would preclude participation in this study or interfere with compliance.
* Current diagnosis of cardiovascular disease, diabetes, or cancer (except for non-melanoma skin cancer).
* History of allergic reactions to blueberries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of inflammasome ASC oligomers | Change from pre-study to post-2 weeks supplementation, and immediately post-exercise, and 1.5 hours-, and 24 hours-post-exercise
  ASC oligomers are an indicator of inflammasome activation

SECONDARY OUTCOMES:
Plasma concentrations of 4-hydroxynonenal | Change from pre-study to post-2 weeks supplementation, and immediately post-exercise, and 1.5 hours-, and 24 hours-post-exercise
  Oxidative stress measure
Urine concentrations of hippuric acid | Change from pre-study to post-2 weeks supplementation, and immediately post-exercise, and 1.5 hours-, and 24 hours-post-exercise
  Blueberry metabolite

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Summer, 2024